CLINICAL TRIAL: NCT05299476
Title: A Single-arm, Open Phase II Trial of CAPOX Combined With Bevacizumab Combined With Tislelizumab in First-line Treatment of PDL1 CPS < 5 Locally Advanced or Metastati Gastroesophageal Adenocarcinoma
Brief Title: CAPOX + Bevacizumab + Tislelizumab Treating PD-L1 CPS < 5 Locally Advanced or Metastatic GEA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dai, Guanghai, Director, Department of Oncology, PLA General Hospital, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2021-642-01
Record Dates: First submitted 2022-03-01; First posted 2022-03-29 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-04

CONDITIONS: Advanced Gastroesophageal Adenocarcinoma; First-line Therapy; PDL1 CPS < 5
MeSH Terms: interventions — Bevacizumab; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAPOX combined with bevacizumab and Tislelizumab (Experimental)
  Interventions: Drug: CAPOX combined with bevacizumab and Tislelizumab

INTERVENTIONS:
Drug: CAPOX combined with bevacizumab and Tislelizumab — Oxaliplatin: intravenous infusion, 130mg/m2, infusion for more than 3h, every 3 weeks for a cycle, infusion 4-8 cycles; Capecitabine: oral administration, 2g/m2, 2 times, 14 days, 7 days rest, every 3 weeks for a cycle; Bevacizumab was administered intravenously (without prophylaxis) at 7.5mg/kg. The first infusion was 90min, the second infusion was 60min, and each infusion was 30 min. The drug was administered once every 3 weeks, and the longest cumulative duration was 2 years.
  Tislelizumab is administered intravenously (without prophylaxis) at a fixed dose of 200mg. Each infusion was 30 min (no less than 20 min, no more than 60 min), and the drug was given once every 3 weeks for a cycle, with the longest cumulative duration of 2 years.

SUMMARY:
his study was a single-arm, open, single-center Phase ii clinical trial to observe and evaluate the efficacy and safety of CAPOX+ bevacizumab + tislelizumab in first-line treatment of ADVANCED gastroesophageal adenocarcinoma with CPS < 5.

This study targeted advanced gastric cancer patients who could not undergo radical treatment, who had not received systemic therapy before, or who had recurrence and metastasis more than 6 months after the end of adjuvant therapy.

The 6-month progression-free survival (PFS) rate will be used as the primary outcome indicator, and approximately 30 subjects will be enrolled.

Subject will receive CAPOX+ bevacizumab + tislelizumab continuously for a treatment cycle of 3 weeks after fully informed and signing informed consent, oxaliplatin will be stopped after 4-8 cycles, and other drugs will continue to be used until the treatment interruption event specified in the plan occurs. Post-treatment follow-up for safety and survival will continue after completion of treatment, and follow-up for tumor progression will also be conducted after completion of treatment for subjects who have not finished treatment for a cause of disease progression/death.

After the subjects were enrolled in the study, safety visits were conducted for each treatment cycle D1 before medication. Imaging will be performed every 2 cycles from the first year of treatment to assess efficacy, and every 3 cycles after 1 year until treatment ends, informed consent is withdrawn, or death.

ELIGIBILITY:
Inclusion Criteria:

* At the same time, patients voluntarily participated in the study and signed informed consent.
* Either male or female, aged 18 or older.
* Patients diagnosed by pathological or cytological diagnosis of gastric cancer (GC), gastroesophageal junction carcinoma (GEJ) or esophageal adenocarcinoma had evidence of local advanced lesions or metastases that could not be surgically resected, and were mostly adenocarcinoma confirmed by histological examination.
* Anyway, she has no previous systemic therapy; Or had received neoadjuvant/adjuvant chemotherapy but experienced disease progression or recurrence 6 months after the end of treatment;
* PDL-1 CPS < 5, HER2 negative;
* Anyway, ECOG scores 0-1 on PS.Estimated survival ≥3 months;
* Anyway, their vital organs function according to the following rules:

  1. Hemoglobin (HGB) ≥90g/L;
  2. Neutrophil count (ANC) ≥1.5×109/L;
  3. Platelet count (PLT) ≥80×109/L;
  4. ALT and AST≤2.5×ULN;ALT and AST≤5×ULN for liver metastasis;
  5. Total bilirubin (TBIL) ≤1.5 times normal upper limit (ULN);
  6. Serum Cr≤1×ULN, endogenous creatinine clearance rate > 50ml/min (Cockcroft-Gault formula);
  7. Urinary protein < (++), or 24-hour urinary protein < 1.0g;
* Lent blood functions normally, without active bleeding or thrombotic disease:

  1. INR≤1.5×ULN;
  2. Partial thrombin time APTT≤1.5×ULN;
  3. Prothrombin time PT≤1.5×ULN;
* Women of reproductive age had to undergo a pregnancy test (serum or urine) which was negative within 7 days of enrollment, and volunteer to use an appropriate method of contraception during the observation period and for 12 weeks after the last study drug was given. For men, surgical sterilization or consent to use appropriate methods of contraception during the observation period and for 12 weeks after the last administration of the study drug;
* Anyway, people who comply are expected to be able to follow up on therapeutic outcomes and adverse reactions as required by the regimen.

Exclusion Criteria:

* Five years before first use of the study drug has been diagnosed as other malignant tumor, the effective treatment of basal cell carcinoma, squamous cell carcinoma of the skin and/or the effective removal of cervical cancer in situ and/or except breast cancer.
* Known allergy to oxaliplatin, PD-1 mab, bevacizumab or pharmaceutical excipients;Or severe allergic reactions to other monoclonal antibodies;
* Chauvinist has any active autoimmune disease or a history of autoimmune disease (e.g. interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis,vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (which can be included after hormone replacement therapy); Patients with complete remission of childhood asthma without intervention or vitiligo as adults may be included, but not those requiring medical intervention with bronchodilators;
* HBV DNA>500 IU/ mL (or 2000 copies /ml), HCV RNA>103 copies /ml, HBsAg+ and anti-HCV antibody positive;
* Lent has a history of HIV infection;
* Accuser spends 14 days prior to first using a study drug, regardless of nasal spray and inhaled corticosteroids or physiological doses of systemic steroids (i.e., no more than 10 mg/ day of prednisone or an equivalent pharmacophysiological dose of another corticosteroid);
* A live attenuated vaccine was administered either four weeks before the first dose or during the study period;
* History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation is known；
* Hypertension that cannot be controlled even with standard treatment (systolic blood pressure ≥160mmHg/ diastolic blood pressure ≥100mmHg);
* Either having poorly controlled cardiac clinical symptoms or disease, such as :(1) NYHA grade 2 or higher heart failure, (2) unstable angina, (3) myocardial infarction within 1 year, or (4) clinically significant supracventricular or ventricular arrhythmias requiring treatment or intervention;
* Patients at risk of serious bleeding, including but not limited to severe bleeding (bleeding > 30 ml within 3 months), were evaluated by a physician who agreed to spend time on an endoscopic evaluation, which was subject to endoscopic evaluation.
* Either a thromboembolic event (including a stroke event and/or a transient ischemic attack) occurs within 6 months;
* Participates in another clinical trial, or participates in any other drug clinical study within four weeks, or at least five half-lives since the last study drug was taken;
* At the same time, participants in the Study underwent anti-tumor therapy including chemotherapy, radiotherapy and immunotherapy within 4 weeks prior to drug administration.
* At the same time, participants received palliative radiotherapy for bone metastasis within 2 weeks prior to the beginning of drug administration. Radiation therapy for other sites within the first 4 weeks;
* Regardless, toxicity from previous anti-tumor therapy does not return to CTCAE [version 5.0] level 0-1, as shown in the following.Except: a. hair loss;B. Pigmentation;C. Long-term toxicity caused by radiotherapy could not be recovered according to the judgment of researchers;
* Other conditions that the investigator deems inappropriate for inclusion;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
6-month progression-free survival | Six months from the start of treatment
  Probability of disease-free progression within 6 months in patients with complete remission and in patients with partial remission or disease progression

SECONDARY OUTCOMES:
ORR（Objective Response Rate） | Imaging tests were performed every 6 weeks (±7 days) from the first year of treatment to assess efficacy, and every 9 weeks (±7 days) after 1 year
  The proportion of patients whose tumors shrink by a certain amount and remain so for a certain amount of time, including CR+PR cases.
PFS（progression-free survival） | Imaging tests were performed every 6 weeks (±7 days) from the first year of treatment to assess efficacy, and every 9 weeks (±7 days) after 1 year
  Time from randomness to the first occurrence of disease progression or death from any cause.
OS（Overall Survival) | Imaging tests were performed every 6 weeks (±7 days) from the first year of treatment to assess efficacy, and every 9 weeks (±7 days) after 1 year
  Time from randomization to death from any cause
Time to Response (TTR) | From enrollment to the end of treatment at 8 weeks
  TTR was defined as the time from randomization to the first occurrence of CR or PR.
Adverse Event | Safety visits were made before medication in each treatment cycle day1(every cycle is 21days)
  The dose suspension rate and dose termination rate caused by adverse events were determined according to NCI-CTCAE V5.0 standard
Duration of Response (DOR) | From enrollment to the end of treatment at 8 weeks
  duration of response (DOR) defined as the period between the first objective response and the first documented PD or death of any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Runge TM, Abrams JA, Shaheen NJ. Epidemiology of Barrett's Esophagus and Esophageal Adenocarcinoma. Gastroenterol Clin North Am. 2015 Jun;44(2):203-31. doi: 10.1016/j.gtc.2015.02.001. Epub 2015 Apr 9. PMID 26021191
- [Background] Hur C, Miller M, Kong CY, Dowling EC, Nattinger KJ, Dunn M, Feuer EJ. Trends in esophageal adenocarcinoma incidence and mortality. Cancer. 2013 Mar 15;119(6):1149-58. doi: 10.1002/cncr.27834. Epub 2012 Dec 11. PMID 23303625
- [Background] Kanat O, O'Neil B, Shahda S. Targeted therapy for advanced gastric cancer: A review of current status and future prospects. World J Gastrointest Oncol. 2015 Dec 15;7(12):401-10. doi: 10.4251/wjgo.v7.i12.401. PMID 26690491
- [Background] De Vita F, Di Martino N, Fabozzi A, Laterza MM, Ventriglia J, Savastano B, Petrillo A, Gambardella V, Sforza V, Marano L, Auricchio A, Galizia G, Ciardiello F, Orditura M. Clinical management of advanced gastric cancer: the role of new molecular drugs. World J Gastroenterol. 2014 Oct 28;20(40):14537-58. doi: 10.3748/wjg.v20.i40.14537. PMID 25356019
- [Background] Orditura M, Galizia G, Sforza V, Gambardella V, Fabozzi A, Laterza MM, Andreozzi F, Ventriglia J, Savastano B, Mabilia A, Lieto E, Ciardiello F, De Vita F. Treatment of gastric cancer. World J Gastroenterol. 2014 Feb 21;20(7):1635-49. doi: 10.3748/wjg.v20.i7.1635. PMID 24587643
- [Background] Janjigian YY, Shitara K, Moehler M, Garrido M, Salman P, Shen L, Wyrwicz L, Yamaguchi K, Skoczylas T, Campos Bragagnoli A, Liu T, Schenker M, Yanez P, Tehfe M, Kowalyszyn R, Karamouzis MV, Bruges R, Zander T, Pazo-Cid R, Hitre E, Feeney K, Cleary JM, Poulart V, Cullen D, Lei M, Xiao H, Kondo K, Li M, Ajani JA. First-line nivolumab plus chemotherapy versus chemotherapy alone for advanced gastric, gastro-oesophageal junction, and oesophageal adenocarcinoma (CheckMate 649): a randomised, open-label, phase 3 trial. Lancet. 2021 Jul 3;398(10294):27-40. doi: 10.1016/S0140-6736(21)00797-2. Epub 2021 Jun 5. PMID 34102137
- [Background] Hagi T, Kurokawa Y, Kawabata R, Omori T, Matsuyama J, Fujitani K, Hirao M, Akamaru Y, Takahashi T, Yamasaki M, Satoh T, Eguchi H, Doki Y. Multicentre biomarker cohort study on the efficacy of nivolumab treatment for gastric cancer. Br J Cancer. 2020 Sep;123(6):965-972. doi: 10.1038/s41416-020-0975-7. Epub 2020 Jul 3. PMID 32616848
- [Background] Boku N, Ryu MH, Kato K, Chung HC, Minashi K, Lee KW, Cho H, Kang WK, Komatsu Y, Tsuda M, Yamaguchi K, Hara H, Fumita S, Azuma M, Chen LT, Kang YK. Safety and efficacy of nivolumab in combination with S-1/capecitabine plus oxaliplatin in patients with previously untreated, unresectable, advanced, or recurrent gastric/gastroesophageal junction cancer: interim results of a randomized, phase II trial (ATTRACTION-4). Ann Oncol. 2019 Feb 1;30(2):250-258. doi: 10.1093/annonc/mdy540. PMID 30566590
- [Background] Friedlander M, Meniawy T, Markman B, Mileshkin L, Harnett P, Millward M, Lundy J, Freimund A, Norris C, Mu S, Wu J, Paton V, Gao B. Pamiparib in combination with tislelizumab in patients with advanced solid tumours: results from the dose-escalation stage of a multicentre, open-label, phase 1a/b trial. Lancet Oncol. 2019 Sep;20(9):1306-1315. doi: 10.1016/S1470-2045(19)30396-1. Epub 2019 Aug 1. PMID 31378459
- [Background] Zhang T, Song X, Xu L, Ma J, Zhang Y, Gong W, Zhang Y, Zhou X, Wang Z, Wang Y, Shi Y, Bai H, Liu N, Yang X, Cui X, Cao Y, Liu Q, Song J, Li Y, Tang Z, Guo M, Wang L, Li K. The binding of an anti-PD-1 antibody to FcgammaRIota has a profound impact on its biological functions. Cancer Immunol Immunother. 2018 Jul;67(7):1079-1090. doi: 10.1007/s00262-018-2160-x. Epub 2018 Apr 23. PMID 29687231
- [Background] Song Y, Gao Q, Zhang H, Fan L, Zhou J, Zou D, Li W, Yang H, Liu T, Wang Q, Lv F, Guo H, Yang L, Elstrom R, Huang J, Novotny W, Wei V, Zhu J. Treatment of relapsed or refractory classical Hodgkin lymphoma with the anti-PD-1, tislelizumab: results of a phase 2, single-arm, multicenter study. Leukemia. 2020 Feb;34(2):533-542. doi: 10.1038/s41375-019-0545-2. Epub 2019 Sep 13. PMID 31520078
- [Background] Desai J, Deva S, Lee JS, Lin CC, Yen CJ, Chao Y, Keam B, Jameson M, Hou MM, Kang YK, Markman B, Lu CH, Rau KM, Lee KH, Horvath L, Friedlander M, Hill A, Sandhu S, Barlow P, Wu CY, Zhang Y, Liang L, Wu J, Paton V, Millward M. Phase IA/IB study of single-agent tislelizumab, an investigational anti-PD-1 antibody, in solid tumors. J Immunother Cancer. 2020 Jun;8(1):e000453. doi: 10.1136/jitc-2019-000453. PMID 32540858
- [Background] Shen L, Guo J, Zhang Q, Pan H, Yuan Y, Bai Y, Liu T, Zhou Q, Zhao J, Shu Y, Huang X, Wang S, Wang J, Zhou A, Ye D, Sun T, Gao Y, Yang S, Wang Z, Li J, Wu YL. Tislelizumab in Chinese patients with advanced solid tumors: an open-label, non-comparative, phase 1/2 study. J Immunother Cancer. 2020 Jun;8(1):e000437. doi: 10.1136/jitc-2019-000437. PMID 32561638
- [Background] Xu J, Bai Y, Xu N, Li E, Wang B, Wang J, Li X, Wang X, Yuan X. Tislelizumab Plus Chemotherapy as First-line Treatment for Advanced Esophageal Squamous Cell Carcinoma and Gastric/Gastroesophageal Junction Adenocarcinoma. Clin Cancer Res. 2020 Sep 1;26(17):4542-4550. doi: 10.1158/1078-0432.CCR-19-3561. Epub 2020 Jun 19. PMID 32561664
- [Background] Van Cutsem E, de Haas S, Kang YK, Ohtsu A, Tebbutt NC, Ming Xu J, Peng Yong W, Langer B, Delmar P, Scherer SJ, Shah MA. Bevacizumab in combination with chemotherapy as first-line therapy in advanced gastric cancer: a biomarker evaluation from the AVAGAST randomized phase III trial. J Clin Oncol. 2012 Jun 10;30(17):2119-27. doi: 10.1200/JCO.2011.39.9824. Epub 2012 May 7. PMID 22565005
- [Background] Wilke H, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Sugimoto N, Lipatov O, Kim TY, Cunningham D, Rougier P, Komatsu Y, Ajani J, Emig M, Carlesi R, Ferry D, Chandrawansa K, Schwartz JD, Ohtsu A; RAINBOW Study Group. Ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (RAINBOW): a double-blind, randomised phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1224-35. doi: 10.1016/S1470-2045(14)70420-6. Epub 2014 Sep 17. PMID 25240821
- [Background] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585
- [Background] Fukuoka S, Hara H, Takahashi N, Kojima T, Kawazoe A, Asayama M, Yoshii T, Kotani D, Tamura H, Mikamoto Y, Hirano N, Wakabayashi M, Nomura S, Sato A, Kuwata T, Togashi Y, Nishikawa H, Shitara K. Regorafenib Plus Nivolumab in Patients With Advanced Gastric or Colorectal Cancer: An Open-Label, Dose-Escalation, and Dose-Expansion Phase Ib Trial (REGONIVO, EPOC1603). J Clin Oncol. 2020 Jun 20;38(18):2053-2061. doi: 10.1200/JCO.19.03296. Epub 2020 Apr 28. PMID 32343640
- [Background] Nakajima TE, Kadowaki S, Minashi K, Nishina T, Yamanaka T, Hayashi Y, Izawa N, Muro K, Hironaka S, Kajiwara T, Kawakami Y. Multicenter Phase I/II Study of Nivolumab Combined with Paclitaxel Plus Ramucirumab as Second-line Treatment in Patients with Advanced Gastric Cancer. Clin Cancer Res. 2021 Feb 15;27(4):1029-1036. doi: 10.1158/1078-0432.CCR-20-3559. Epub 2020 Dec 1. PMID 33262133
- [Background] Chu T, Lu J, Bi M, Zhang H, Zhuang W, Yu Y, Shi J, Chen Z, Zhang X, Guo Q, Liu Q, Wu H, Fang J, Hu Y, Wang X, Han C, Li K, Han B. Equivalent efficacy study of QL1101 and bevacizumab on untreated advanced non-squamous non-small cell lung cancer patients: a phase 3 randomized, double-blind clinical trial. Cancer Biol Med. 2021 Mar 12;18(3):816-24. doi: 10.20892/j.issn.2095-3941.2020.0212. PMID 33710815
- See also: Related Info — http://clinicaltrials.gov/ct2/show/NCT03777657.